CLINICAL TRIAL: NCT05902949
Title: Analysis of Postural Control in Children After of Exercise Therapy Versus Passive "Heel Pad" Treatment: Randomized Controlled Trial.
Brief Title: Analysis of Postural Control in Children Suffering From Triceps Suralis Shortening.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCV/2017-2018//113
Record Dates: First submitted 2022-11-29; First posted 2023-06-15 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Ankle Disease
Keywords: Muscle Stretching Exercises; Balance; Exercise; Range of Motion
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching Group (Active Comparator): The pattern will be performed 3 times per day (10 repetitions, 30 seconds each repetition). A daily control diary will be filled in when performing the exercise.
  Interventions: Procedure: Streching Group
- Heel Cup Group (Active Comparator): The heel cup will be 5mm high (Eva Shore 65)
  Interventions: Procedure: Heel group

INTERVENTIONS:
Procedure: Streching Group — The Streching group will perform a conventional stretching exercise.
  Arms: Stretching Group
Procedure: Heel group — The heel pad group will be applied a plantar support during the months of the study.
  Arms: Heel Cup Group

SUMMARY:
The central nervous system (CNS) coordinates balance through the visual, vestibular, and somatoproprioceptive systems, which produce muscle activation for postural control. Among the important muscle activations for postural control are those produced in the ankle joint, which is crucial for maintaining postural control in sports settings, along with the gastrocnemius and soleus muscles. Studies show that children who practice sports improve their postural stability and accelerate sensory maturation, which can affect the development of the lower limb extremity, specifically the insertional musculature of the ankle and foot. The present study aims to analyze postural control in school-aged children with triceps suralis retraction and assess the effectiveness of treatment with stretching versus a heel pad for 3 and 6 months. Additionally, the study will analyze whether the physical activity the children engage in influences their stability

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted to evaluate the effectiveness of using a heel pad and a gastrocnemius and soleus stretching protocol. The outcomes of both interventions will be evaluated and compared, including pre-intervention and post-intervention assessments at 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Children 8-12 years old
2. Regular sports practice
3. Decreased range of flexión

Exclusion Criteria:

1. Having neurological, vestibular, muscular, psychological or visual visual disease.
2. Traumatic pathology 12 months prior to the measurement (sprains, talalgias, etc.).
3. Diseases of balance or motor control.
4. Surgeries in the last 12 months.
5. Taking medications that may affect the neuromuscular system.
6. Sports practice in the last 48 hours.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Physical Activity Questionnaire for Children (PAQ-C) at 6 months | At baseline; post 1 (3 months) and post 2 (6 months)
  The data on the type and amount of physical activity performed by the participants will be collected using the Spanish version of the Physical Activity Questionnaire for Children (PAQ-C) (Appendix 3). The PAQ-C has been validated by Manchola-González, Bagur-Calafat, and Girabent-Farrésby Manchola-González, Bagur-Calafat, and Girabent-Farrés will be used to collect data on the type and amount of physical activity performed by the participants.

SECONDARY OUTCOMES:
Stabilometry | At baseline; post 1 (3 months) and post 2 (6 months)
  For collecting stabilometry data, an inertial measurement instrument called Gyko® (Janusz Jaworski et al., 2020) (Figure 5) will be used. It is a state-of-the-art device that allows for objective assessment of acceleration, angular velocity, and with an acquisition frequency of 100Hz
Instability test | At baseline; post 1 (3 months) and post 2 (6 months)
  The instability test will be performed using a foam rubber pad model Balance _Pand Elite ® with dimensions of 50 x 41 x 6cm, a weight of 0.7kg, and a density of 55kg/m (Figure 6). The foam has a nominal density of 40kg/m3 and a vertical compressive strength of 0.45N mm2 and a vertical compressive elasticity of 34N mm2 according to the manufacturer
Lunge Test | At baseline; post 1 (3 months) and post 2 (6 months)
  he Lunge Test will be used to determine the dorsal flexion of the ankle (Figure 10) using the Leg MOtion® system

CONTACTS AND LOCATIONS:
Locations (1):
- Javier Ferrer Torregrosa, Torrent, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Soidan JL, Garcia-Lineira J, Leiros-Rodriguez R, Soto-Rodriguez A. Physical Activity Practice and Optimal Development of Postural Control in School Children: Are They Related? J Clin Med. 2020 Sep 10;9(9):2919. doi: 10.3390/jcm9092919. PMID 32927763
- [Background] Vallandingham RA, Gaven SL, Powden CJ. Changes in Dorsiflexion and Dynamic Postural Control After Mobilizations in Individuals With Chronic Ankle Instability: A Systematic Review and Meta-Analysis. J Athl Train. 2019 Apr;54(4):403-417. doi: 10.4085/1062-6050-380-17. Epub 2019 Mar 14. PMID 30870009
- [Background] Martinez-Corcoles V, Nieto-Gil P, Ramos-Petersen L, Ferrer-Torregrosa J. Balance performance analysis after the COVID-19 quarantine in children aged between 8 and 12 years old: Longitudinal study. Gait Posture. 2022 May;94:203-209. doi: 10.1016/j.gaitpost.2022.03.019. Epub 2022 Mar 27. PMID 35366430
- [Background] Hsu YS, Kuan CC, Young YH. Assessing the development of balance function in children using stabilometry. Int J Pediatr Otorhinolaryngol. 2009 May;73(5):737-40. doi: 10.1016/j.ijporl.2009.01.016. Epub 2009 Feb 20. PMID 19232750
- [Background] Hoch MC, Staton GS, McKeon PO. Dorsiflexion range of motion significantly influences dynamic balance. J Sci Med Sport. 2011 Jan;14(1):90-2. doi: 10.1016/j.jsams.2010.08.001. Epub 2010 Sep 16. PMID 20843744
- [Background] Han J, Anson J, Waddington G, Adams R, Liu Y. The Role of Ankle Proprioception for Balance Control in relation to Sports Performance and Injury. Biomed Res Int. 2015;2015:842804. doi: 10.1155/2015/842804. Epub 2015 Oct 25. PMID 26583139
- [Background] Grindstaff TL, Dolan N, Morton SK. Ankle dorsiflexion range of motion influences Lateral Step Down Test scores in individuals with chronic ankle instability. Phys Ther Sport. 2017 Jan;23:75-81. doi: 10.1016/j.ptsp.2016.07.008. Epub 2016 Jul 29. PMID 27662790
- [Derived] Martinez-Corcoles V, Garcia-Campos J, Vicente-Mampel J, Chicharro-Luna E, Jimenez EMM, Ferrer-Torregrosa J. Postural analysis of children with muscle retraction after six-month exercise or heel cup interventions in a randomized trial. Sci Rep. 2025 Apr 19;15(1):13578. doi: 10.1038/s41598-025-98527-6. PMID 40253482